CLINICAL TRIAL: NCT03640754
Title: Study to Assess the Safety and Effect of Repeated Administration of Granulocyte Colony-Stimulating Factor (G-CSF; Filgrastim) on Hot Flashes and Other Vasomotor Symptoms of Menopause in Postmenopausal Women
Brief Title: A Study of the Safety and Effect of Repeated Administration of G-CSF on Hot Flashes in Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MenoGeniX, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MNGX-102; 1R43AG056209-01A1 (NIH)
Record Dates: First submitted 2018-07-30; First posted 2018-08-21 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Postmenopausal Symptoms
Keywords: Hot Flashes; Vasomotor Symptoms; Menopause
MeSH Terms: conditions — Hot Flashes | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental: G-CSF (Active Comparator): Intervention: G-CSF given by subcutaneous injection repeated 3 times (Days 0, 28, 56) Other name: Filgrastim
  Interventions: Biological: G-CSF
- Comparator: Placebo/Saline (Placebo Comparator): Intervention: Placebo/saline given by subcutaneous injection repeated 3 times (Days 0, 28, 56) Other name: Saline
  Interventions: Other: Placebo/Saline

INTERVENTIONS:
Biological: G-CSF — G-CSF injected subcutaneously 3 times (Days 0, 28, 56)
  Other Names: Filgrastim
  Arms: Experimental: G-CSF
Other: Placebo/Saline — Placebo/saline injected subcutaneously 3 times (Days 0, 28, 56)
  Other Names: Saline
  Arms: Comparator: Placebo/Saline

SUMMARY:
The purpose of this study is to assess the efficacy and safety of repeated administration of G-CSF for the treatment of hot flashes and vasomotor symptoms in women with naturally-occurring or surgically induced menopause. G-CSF will be administered three times at 28 day intervals to postmenopausal women, ages 40 to 65, suffering at least 49 moderate to severe hot flashes per week.

DETAILED DESCRIPTION:
This is a 12-week, multicenter, randomized, double-blind, placebo-controlled study. Eligible subjects will be stratified by natural or surgical menopause and randomized (1:1) to receive 3 single injections, 28-days apart, of either G-CSF or placebo.

This study will consist of a 14-21 day screening period. Subjects enrolled will be given three single 1.0 mL subcutaneous (SC) injections (repeated 28-days apart), in the outer area of either upper arm, of either G-CSF or placebo (sterile physiological saline) at Baseline, Day 28 and Day 56. Subjects will be followed for 12 weeks and will complete hot flash diary entries every day for the duration of treatment. Safety will be assessed by adverse events, clinical laboratory tests (clinical chemistry and complete blood count with differential) and vital signs. A follow-up phone call will occur 60 days after the last dose of study drug.

Eligibility will be assessed via physical examination, clinical laboratory testing, vital signs.

Subjects will receive a diary in which to record daily hot flashes symptoms during the duration of the screening period. Subjects must have at least 14 days of hot flash recordings to participate in the study. The diary will be reviewed by study site staff on Baseline (Day 0) to confirm study eligibility.

During the treatment period, subjects will return to the study site at Days 1, 21, 28, 29, 49, 56, 57, and 84 for assessments.

The follow-up phone call will occur approximately 60 days following the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 49 to 65 for natural postmenopausal or aged 40 to 65 for surgical postmenopausal
* Body Mass Index (BMI) 18 to 35
* At least 7 moderate to severe hot flashes per day on average (or at least 49 moderate to severe hot flashes per week)
* Naturally postmenopausal or surgically postmenopausal women:
* Naturally postmenopausal is defined as having no menstrual periods for at least 12 months prior to study entry; with a biochemical criteria of menopause (FSH >40 IU/L)
* Surgically postmenopausal is defined as at least 3 months after documented bilateral salpingo oophorectomy
* Normal pelvic exam and pap smear within 2 years
* Signed informed consent

Exclusion Criteria:

* Radiation or chemotherapy-induced (including gonadotropin-releasing hormone (GnRH) agonist) menopause
* Prior chemotherapy or radiation therapy for cancer
* Prior diagnosis of hematologic malignancy
* Type 1 diabetics or Type 2 diabetics with HbA1c > 7.0%
* Use of hormone replacement therapy or oral contraceptives within the past three months
* Use of alternative or complementary medicines or herbs for menopausal symptoms within 30 days (refer to Appendix 2)
* Use of any selective serotonin reuptake inhibitor (SSRI) or serotonin norepinephrine reuptake inhibitor (SNRI) within 30 days
* Use of selective estrogen receptor modulators within 30 days
* Use of gabapentin within 30 days
* Use of clonidine within 30 days
* Use of megestrol acetate (Megace) within 30 days
* Use of, prescription corticosteroids within 30 days (nasal or other inhaled corticosteroids and over-the-counter (OTC) hydrocortisone ointment or cream excepted)
* Current use of lithium therapy (related to possible risk of G-CSF)
* History (in the past year) or presence of drug or alcohol use which, in the opinion of the Investigator, might compromise the study or confound the study results
* History of use of any anti-inflammatory biologics
* History of or current splenomegaly (related to possible risk of G-CSF)
* History of sickle cell disease (related to possible risk of G-CSF)
* High risk for medical complications that might affect the subject's ability to complete the trial without a serious co-morbid event, based on medical history, physical examination and laboratory screening evaluation in the opinion of the Investigator
* Presence of an acute or chronic condition (such as a hematological, rheumatologic auto-immune disease, chronic inflammatory disorder or osteoporosis) based on history, clinical, or laboratory evaluation, which, in the opinion of the Investigator, might compromise the study, confound the study results or place the subject at risk
* Follicle stimulating hormone (FSH) < 40 IU/L or below the reference range for menopause for the local laboratory used for screening
* Thyroid stimulating hormone (TSH) outside normal limits at study entry
* Absolute neutrophil count (ANC) ≤ 1.0 x 109/L
* Total white blood cell count (WBC) ≤ 3.0 x 109/L
* Platelet count (PLT) ≤ 150 x 109/L
* Hemoglobin count (HGB) consistent with anemia
* Positive urine pregnancy test at Baseline visit
* Allergy or hypersensitivity to E coli-derived proteins' G-CSF' or any component of the product
* Mentally or legally incapacitated such that informed consent cannot be obtained
* Inability or unwillingness to complete daily hot flash diary and study questionnaires appropriately
* Participation in another investigational trial within the past 30 days

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard C Duke, PhD, Study Chair — MenoGeniX, Inc.
Locations (2):
- United States (2):
  - Site 2, Aurora, Colorado
  - Site 1, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal women participants 40 to 65 years of age who had moderate to severe vasomotor symptoms (VMS) and seeking treatment or relief for hot flashes associated with menopause, confirmed as menopausal, had to have 7 to 8 moderate to severe hot flashes per day within the 7 days prior to randomization and who met the inclusion criteria and none of the exclusion criteria were enrolled in this study. A total of 61 subjects were randomized to receive G-CSF or saline in this trial.
Pre-assignment Details: Prior to randomization, participants had a screening period during which a minimum 7-day collection of baseline hot flash frequency and severity assessments were performed.
Groups:
- Experimental: G-CSF (All Subjects): Intervention: G-CSF (300 mcg/injection as filgrastim) given by subcutaneous injection on days 0, 28 and 56. This group is all women in the study that received G-CSF.
- Comparator: Placebo/Saline (All Subjects): Intervention: Placebo (as saline) given by subcutaneous injection on days 0, 28 and 56. This group is all women in the study that received placebo.
Period: Overall Study
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects)
Started | 31 | 30
Completed | 30 | 29
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental: G-CSF (All Subjects): Intervention: G-CSF given by subcutaneous injection repeated 3 times (Days 0, 28, 56) Other name: Filgrastim
  G-CSF: G-CSF injected subcutaneously 3 times (Days 0, 28, 56)
- Comparator: Placebo/Saline (All Subjects): Intervention: Placebo/saline given by subcutaneous injection repeated 3 times (Days 0, 28, 56) Other name: Saline
  Placebo/Saline: Placebo/saline injected subcutaneously 3 times (Days 0, 28, 56)
- Total: Total of all reporting groups
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] — All randomized participants
  years | 55.4 (4.39) | 55.6 (4.58) | 55.5 (4.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 22 | 23 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Daily Moderate + Severe Hot Flashes (M+S) [Mean (Standard Deviation); unit: Number of hot flashes per day] — Average number of daily moderate (M) and severe (S) hot flashes (M+S) during the seven days prior to randomization to receive G-CSF or placebo.A daily frequency per week was derived by taking the mean of the data over 7 days.
  Number of hot flashes per day | 12.5 (5.14) | 12.3 (4.73) | 12.4 (4.9)
Composite Daily Hot Flash Severity (CDS) [Mean (Standard Deviation); unit: Number of hot flashes per day] — CDS = (number of daily mild hot flashes x1) + (number of daily moderate hot flashes x2) + (number of severe hot flashes x3) during the seven days preceding randomization. A daily frequency per week was derived by taking the mean of the data over 7 days.
  Number of hot flashes per day | 33.7 (12.72) | 33.7 (14.44) | 33.7 (13.49)
Hot Flash Severity Score (HFSS) [Mean (Standard Deviation); unit: Score on a scale] — HFSS = ((number of daily mild hot flashes x1) + (number of daily moderate hot flashes x2) + (number of severe hot flashes x3))/daily total hot flashes) during the seven days preceding randomization, where total hot flashes (THF) = number of daily mild, moderate, and severe hot flashes during the seven days prior to randomization. A daily frequency per week was derived by taking the mean of the data over 7 days.
  Score on a scale | 2.3 (0.32) | 2.4 (0.35) | 2.3 (0.34)
White Blood Cell Counts (WBC) [Mean (Standard Deviation); unit: White Blood Cells per mL] — Blood samples were obtained on day 0 upon randomization and first administration of G-CSF or placebo.
  White Blood Cells per mL | 6007 (1923) | 6142 (1296) | 6088 (1633)
Menopause-specific Quality of Life Questionnaire - Vasomotor symptom (MENQOL VMS) Score [Mean (Standard Deviation); unit: Score on a scale] — Menopause-specific Quality of Life (MENQOL) Questionnaire. The MENQOL is self-administered and consists of a total of 29 items in a Likert-scale format. Each item assesses the impact of one of four domains of menopausal symptoms, as experienced over the last month: vasomotor (items 1-3), psychosocial (items 4-10), physical (items 11-26), and sexual (items 27-29). MENQOL VMS refers to the answers to items 1-3 where 6 = most bothersome and 0 = least bothersome). (Maximum bother = 18; No bother = 0)
  Score on a scale | 15.5 (2.6) | 15.6 (2.5) | 15.6 (2.5)
Hot Flash Related Daily Interference Scale (HFRDIS) Score [Mean (Standard Deviation); unit: Score on a scale] — The Hot Flash Related Daily Interference Scale (HFRDIS) measures (as a score of 0 to 10) the effect of hot flashes on overall quality of life and on nine specific activities: work, social activities, leisure activities, sleep, mood, concentration, relations with others, sexuality, and enjoyment of life. The 10 answers are added up to get a total score.HFRDIS Score (Maximum Bother = 100; No Bother = 0). The higher the score, the more bothersome the symptoms.
  Score on a scale | 56.9 (21.5) | 62.6 (18.7) | 59.8 (20.2)
Insomnia Severity Index (ISI) Score [Mean (Standard Deviation); unit: Score on a scale] — The Insomnia Severity Index has seven questions.For each question, most bothersome = 4; not botherrsome = 0. The seven answers are added up to get a total score. Total score categories: 0-7 = No clinically significant insomnia; 8-14 = Subthreshold insomnia; 15-21 = Clinical insomnia (moderate severity); 22-28 = Clinical insomnia (severe)
  Score on a scale | 18.8 (5.1) | 19.4 (5.4) | 19.1 (5.2)
Fatigue Severity Scale (FSS) Score [Mean (Standard Deviation); unit: Score on a scale] — Fatigue Severity Scale (FSS) of Sleep Disorders. The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue. The FSS is a short questionnaire that requires the subject to rate level of fatigue. The FSS questionnaire contains nine statements that rate the severity of fatigue symptoms.Each statement is read and the corresponding number from 1 to 7 is circled. A low value (e.g., 1) indicates strong disagreement with the statement, whereas a high value (e.g., 7) indicates strong agreement. (Maximum bother = 70; No bother = 0)
  Score on a scale | 33.8 (15.6) | 34.0 (15.8) | 33.9 (15.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence, including the exacerbation of a pre-existing condition, in a subject or clinical investigation subject administered a pharmaceutical product. This does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) is any experience that suggests a significant hazard, contraindication, side effect, or precaution. This includes any experience that results in death; is acutely life-threatening; requires inpatient hospitalization or prolongs the existing hospitalization; results in persistent or significant incapacity or substantial disruption of ability to conduct normal life functions; is a congenital anomaly/birth defect; or requires medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: From first dose date up to 30 days after last dose (up to 16 weeks)
Measure: Number; unit: Participants
Groups:
- Experimental: G-CSF (White, NH Subgroup): Intervention: G-CSF (300 mcg/injection as filgrastim) given by subcutaneous injection on days 0, 28 and 56. This is a subgroup of the women in the study that received G-CSF and that self-identified as white, non-Hispanic.
- Comparator: Placebo/Saline (White, NH Subgroup): Intervention: Placebo (as saline) given by subcutaneous injection on days 0, 28 and 56. This is a subgroup of the women in the study that received placebo and that self-identified as white, non-Hispanic.
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Participants
  Treatment Emergent Adverse Events (TEAE) | 24 | 20 | 12 | 10
  Drug-related TEAE | 12 | 3 | 5 | 3
  Serious TEAE | 0 | 0 | 0 | 0
  Drug-related serious TEAE | 0 | 0 | 0 | 0
  TEAE leading to death | 0 | 0 | 0 | 0
  TEAE leading to withdrawal of treatment | 0 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in White Blood Cell Counts 24 Hours After Administration of G-CSF or Placebo on Day 0
Description: Change from baseline in white blood cell counts 24 hours after administration of G-CSF or placebo on day 0. Blood samples were collected 24 hours after adminstration of G-CSF on day 0.
Time Frame: Baseline and day 1
Measure: Mean (Standard Error); unit: Number of white blood cells per mL
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Number of white blood cells per mL | 17493 (822) | 103 (144) | 17394 (1095) | 144 (210)
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); Test type: Superiority; p < 0.001, t-test, 1 sided

3. Primary Outcome: Change From Baseline in White Blood Cell Counts 24 Hours After Administration of G-CSF or Placebo on Day 28
Description: Change from baseline in white blood cell counts 24 hours after administration of G-CSF or placebo on day 28. Blood samples were collected 24 hours after adminstration of G-CSF on day 28.
Time Frame: Baseline and day 29
Measure: Mean (Standard Error); unit: Number of white blood cells per mL
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Number of white blood cells per mL | 18273 (988) | 13 (182) | 18378 (1147) | 67 (230)
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); Test type: Superiority; p < 0.001, t-test, 1 sided

4. Primary Outcome: Change From Baseline in White Blood Cell Counts 24 Hours After Administration of G-CSF or Placebo on Day 56.
Description: Change from baseline in white blood cell counts 24 hours after administration of G-CSF or placebo on day 56. Blood samples were collected 24 hours after adminstration of G-CSF on day 56.
Time Frame: Baseline and day 57
Measure: Mean (Standard Error); unit: Number of white blood cells per mL
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Number of white blood cells per mL | 16403 (1445) | 37 (208) | 15128 (2112) | 150 (340)
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); Test type: Superiority; p < 0.001, t-test, 1 sided

5. Primary Outcome: Change From Baseline in White Blood Cell Counts on Day 84 (28 Days After Last Administration of G-CSF or Palcebo)
Description: Change from baseline in white blood cell counts on day 84. Blood samples were collected 24 hours after adminstration of G-CSF on day 84.
Time Frame: Baseline and day 84
Measure: Mean (Standard Error); unit: Number of white blood cells per mL
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Number of white blood cells per mL | -107 (311) | -420 (311) | -611 (297) | -256 (265)
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Test type: Superiority; p = 0.199, t-test, 1 sided
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); Test type: Superiority; p = 0.189, t-test, 1 sided

6. Primary Outcome: Change From Baseline in the Mean Frequency of Moderate and Severe (M+S) Hot Flashes at Week 4
Description: The frequency of moderate to severe hot flashes was the number of moderate to severe hot flashes per 24 hours. A daily frequency per week was derived by taking the mean of the data over 7 days. All subjects who were randomized and received at least one dose of study drug are included in this subset. Subjects are analysed according to the randomized treatment group regardless of treatment received.
Time Frame: Baseline and week 4
Population: Full analysis set (FAS) (consisted of all randomized participants who took at least 1 dose of study intervention) with available data at specified time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of hot flashes per day
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Number of hot flashes per day | -3.9 [-5.7 to -2.2] | -4.0 [-5.7 to -2.3] | -4.1 [-6.4 to -1.8] | -4.0 [-6.2 to -1.7]
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Test type: Superiority — Least squares means (LS Means) from a mixed effects repeated measures model with baseline M+S score, current smoking status, bmi, and parity as covariates; p = 0.398, Mixed Models Analysis
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); Test type: Superiority — [test comment as in outcome 6, analysis 1]; p = 0.391, Mixed Models Analysis

7. Primary Outcome: Change From Baseline in the Mean Frequency of Moderate and Severe (M+S) Hot Flashes at Week 12
Description: as for outcome 6
Time Frame: Baseline and week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of hot flashes per day
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Number of hot flashes per day | -6.4 [-8.2 to -4.7] | -6.0 [-7.7 to -4.3] | -7.5 [-9.9 to -4.3] | -4.5 [-6.8 to -2.2]
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Least squares means (LS Means) from a mixed effects repeated measures model with baseline M+S score, current smoking status, bmi, and parity as covariates; Test type: Superiority; p = 0.232, Mixed Models Analysis
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.085, Mixed Models Analysis

8. Primary Outcome: Change From Baseline in the Mean Composite Daily Severity of Hot Flashes (CDS) at Week 4
Description: CDS (Composite Daily Hot Flash Severity) was calculated as follows:
  [(number of mild hot flashes per day x 1) + (number of moderate hot flashes per day x 2) + (number of severe hot flashes per day x 3)]. A daily frequency per week was derived by taking the mean of the data over 7 days. All subjects who were randomized and received at least one dose of study drug are included in this subset. Subjects are analysed according to the randomized treatment group regardless of treatment received.
Time Frame: Baseline and week 4
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of hot flashes per day
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Number of hot flashes per day | -10 [-15 to -5.5] | -11 [-15 to -6.2] | -11 [-17 to -4.3] | -10 [-17 to -4.3]
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Test type: Superiority; p = 0.501, Mixed Models Analysis
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); Test type: Superiority; p = 0.370, Mixed Models Analysis

9. Primary Outcome: Change From Baseline in the Mean Composite Daily Severity of Hot Flashes (CDS) at Week 12
Description: as for outcome 8
Time Frame: Baseline and week 12
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of hot flashes per day
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Number of hot flashes per day | -17 [-22 to -12] | -16 [-21 to -12] | -19 [-25 to -13] | -12 [-18 to -5.4]
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Test type: Superiority; p = 0.333, Mixed Models Analysis
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); Test type: Superiority; p = 0.014, Mixed Models Analysis

10. Primary Outcome: Change From Baseline in the Mean Daily Severity of Hot Flashes (HFSS) at Week 4
Description: HFSS (Daily Hot Flash Severity Score) was calculated as follows:
  [(number of mild hot flashes per day x 1) + (number of moderate hot flashes per day x 2) + (number of severe hot flashes per day x 3)]/daily total hot flashes), where total hot flashes (THF) = number of daily mild, moderate, and severe hot flashes. A daily severity score per week was derived by taking the mean of the data over 7 days. All subjects who were randomized and received at least one dose of study drug are included in this subset. Subjects are analysed according to the randomized treatment group regardless of treatment received.
Time Frame: Baseline and week 4
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Hot flash severity score
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Hot flash severity score | -0.09 [-0.31 to 0.13] | -0.08 [-0.31 to 0.13] | -0.11 [-0.47 to 0.24] | -0.07 [-0.42 to 0.28]
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Test type: Superiority; p = 0.124, Mixed Models Analysis
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); Test type: Superiority; p = 0.175, Mixed Models Analysis

11. Primary Outcome: Change From Baseline in the Mean Daily Severity of Hot Flashes (HFSS) at Week 12
Description: as for outcome 10
Time Frame: Baseline and week 12
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Hot flash severity score
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Hot flash severity score | -0.31 [-0.53 to -0.09] | -0.13 [-0.34 to 0.09] | -0.43 [-0.79 to -0.08] | -0.19 [-0.55 to 0.17]
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Test type: Superiority; p = 0.032, Mixed Models Analysis
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); Test type: Superiority; p = 0.077, Mixed Models Analysis

12. Secondary Outcome: Number of Subjects Achieving >50% Reduction in the Mean Frequency of Moderate and Severe (M+S) Hot Flashes up to Week 12
Description: as for outcome 6
Time Frame: Weeks 1-12
Population: Full analysis set (FAS) (consisted of all randomized participants who took at least 1 dose of study intervention) with available data at specified time point.
  Outcome Measure Data Table * Measure Type: Least Squares Mean
  * Measure ofDispersion
Measure: Number; unit: Number of subjects
Groups:
- Comparator: Placebo/Saline (White, NH Subgroup): ntervention: Placebo (as saline) given by subcutaneous injection on days 0, 28 and 56. This is a subgroup of the women in the study that received placebo and that self-identified as white, non-Hispanic.
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Number of subjects
  Week 1 | 5 | 4 | 2 | 3
  Week 2 | 8 | 7 | 5 | 3
  Week 3 | 7 | 9 | 5 | 4
  Week 4 | 8 | 8 | 5 | 4
  Week 5 | 15 | 9 | 10 | 3
  Week 6 | 15 | 12 | 10 | 5
  Week 7 | 15 | 12 | 10 | 5
  Week 8 | 12 | 13 | 7 | 5
  Week 9 | 15 | 10 | 9 | 4
  Week 10 | 14 | 12 | 9 | 5
  Week 11 | 15 | 13 | 9 | 6
  Week 12 | 15 | 14 | 9 | 6

13. Secondary Outcome: Number of Subjects Acheiving >50% Reduction in the Mean Composite Daily Hot Flash Severity (CDS) up to Week 12
Description: CDS was calculated as follows:
  [(number of mild hot flashes per day x 1) + (number of moderate hot flashes per day x 2) + (number of severe hot flashes per day x 3)]. A daily frequency per week was derived by taking the mean of the data over 7 days. All subjects who were randomized and received at least one dose of study drug are included in this subset. Subjects are analysed according to the randomized treatment group regardless of treatment received.
Time Frame: Weeks 1-12
Population: as for outcome 6
Measure: Number; unit: Number of subjects
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Number of subjects
  Week 1 | 5 | 4 | 2 | 3
  Week 2 | 8 | 7 | 5 | 3
  Week 3 | 7 | 8 | 5 | 4
  Week 4 | 7 | 7 | 4 | 4
  Week 5 | 15 | 9 | 10 | 3
  Week 6 | 14 | 13 | 10 | 6
  Week 7 | 15 | 11 | 10 | 5
  Week 8 | 12 | 11 | 7 | 4
  Week 9 | 14 | 11 | 8 | 5
  Week 10 | 13 | 12 | 8 | 5
  Week 11 | 15 | 13 | 9 | 6
  Week 12 | 15 | 13 | 9 | 5

14. Secondary Outcome: Number of Subjects Acheiving >0.30 Reduction in the Mean Daily Hot Flash Severity Score (HFSS) up to Week 12
Description: HFSS was calculated as follows:
  [(number of mild hot flashes per day x 1) + (number of moderate hot flashes per day x 2) + (number of severe hot flashes per day x 3)]. HFSS = ((number of daily mild hot flashes x1) + (number of daily moderate hot flashes x2) + (number of severe hot flashes x3))/daily total hot flashes), where total hot flashes (THF) = number of daily mild, moderate, and severe (S) hot flashes. A daily severity score per week was derived by taking the mean of the data over 7 days. All subjects who were randomized and received at least one dose of study drug are included in this subset. Subjects are analysed according to the randomized treatment group regardless of treatment received.
  Severity was zero for participants that had no mild or moderate or severe VMS. Higher scores indicates greater severity.
Time Frame: Weeks 1-12
Population: as for outcome 6
Measure: Number; unit: Number of subjects
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 30 | 18 | 18
Number of subjects
  Week 1 | 4 | 4 | 2 | 3
  Week 2 | 4 | 5 | 3 | 2
  Week 3 | 7 | 6 | 4 | 4
  Week 4 | 5 | 6 | 3 | 4
  Week 5 | 6 | 6 | 3 | 4
  Week 6 | 8 | 5 | 6 | 3
  Week 7 | 7 | 6 | 5 | 4
  Week 8 | 7 | 6 | 5 | 4
  Week 9 | 9 | 5 | 7 | 3
  Week 10 | 8 | 4 | 6 | 2
  Week 11 | 9 | 5 | 6 | 3
  Week 12 | 7 | 6 | 6 | 3

15. Secondary Outcome: Percent Change in M+S at 12 Weeks in Demographic Subgroups
Description: as for outcome 6
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Percent change in hot flashes
Groups:
- Experimental: G-CSF (White, Not Hispanic Subjects): Intervention: G-CSF (300 mcg/injection as filgrastim) given by subcutaneous injection on days 0, 28 and 56. This is a subgroup of the women in the study that received G-CSF and that self-identified as white, non-Hispanic.
- Comparator: Placebo (White, Not Hispanic Subjects): Intervention: Placebo (as saline) given by subcutaneous injection on days 0, 28 and 56. This is a subgroup of the women in the study that received placebo and that self-identified as white, non-Hispanic.
- Experimental: G-CSF (Hispanic Subjects): Intervention: G-CSF (300 mcg/injection as filgrastim) given by subcutaneous injection on days 0, 28 and 56. This is a subgroup of the women in the study that received G-CSF and that self-identified as Hispanic.
- Comparator: Placebo (Hispanic Subjects): Intervention: Placebo (as saline) given by subcutaneous injection on days 0, 28 and 56. This is a subgroup of the women in the study that received placebo and that self-identified as Hispanic.
- Experimental: G-CSF (Black Subjects): Intervention: G-CSF (300 mcg/injection as filgrastim) given by subcutaneous injection on days 0, 28 and 56. This is a subgroup of the women in the study that received G-CSF and that self-identified as Black.
- Comparator: Placebo (Black Subjects): Intervention: Placebo (as saline) given by subcutaneous injection on days 0, 28 and 56. This is a subgroup of the women in the study that received placebo and that self-identified as Black.
Arm/Group | Experimental: G-CSF (White, Not Hispanic Subjects) | Comparator: Placebo (White, Not Hispanic Subjects) | Experimental: G-CSF (Hispanic Subjects) | Comparator: Placebo (Hispanic Subjects) | Experimental: G-CSF (Black Subjects) | Comparator: Placebo (Black Subjects)
Number analyzed (Participants) | 18 | 18 | 6 | 5 | 6 | 6
Percent change in hot flashes | -51 (8) | -33 (8) | -32 (18) | -62 (15) | -46 (18) | -55 (14)
Statistical Analysis 1: Comparison: Experimental: G-CSF (White, Not Hispanic Subjects) vs Comparator: Placebo (White, Not Hispanic Subjects); Test type: Superiority; p = 0.047, t-test, 1 sided
Statistical Analysis 2: Comparison: Experimental: G-CSF (Hispanic Subjects) vs Comparator: Placebo (Hispanic Subjects); Test type: Superiority; p = 0.139, t-test, 1 sided
Statistical Analysis 3: Comparison: Experimental: G-CSF (Black Subjects) vs Comparator: Placebo (Black Subjects); Test type: Superiority; p = 0.395, t-test, 1 sided

16. Secondary Outcome: Net Change in HFSS at 12 Weeks in Demographic Subgroups
Description: HFSS (Daily Hot Flash Severity Score) was calculated as follows:
  [(number of mild hot flashes per day x 1) + (number of moderate hot flashes per day x 2) + (number of severe hot flashes per day x 3)]. HFSS = ((number of daily mild hot flashes x1) + (number of daily moderate hot flashes x2) + (number of severe hot flashes x3))/daily total hot flashes), where total hot flashes (THF) = number of daily mild, moderate, and severe (S) hot flashes. A daily severity score per week was derived by taking the mean of the data over 7 days. All subjects who were randomized and received at least one dose of study drug are included in this subset. Subjects are analysed according to the randomized treatment group regardless of treatment received
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Hot flash severity score
Groups:
- Experimental: G-CSF (White Subjects): Intervention: G-CSF (300 mcg/injection as filgrastim) given by subcutaneous injection on days 0, 28 and 56. This is a subgroup of the women in the study that received G-CSF and that self-identified as white, non-Hispanic.
- Comparator: Placebo (White Subjects): Intervention: Placebo (as saline) given by subcutaneous injection on days 0, 28 and 56. This is a subgroup of the women in the study that received placebo and that self-identified as white, non-Hispanic.
Arm/Group | Experimental: G-CSF (White Subjects) | Comparator: Placebo (White Subjects) | Experimental: G-CSF (Hispanic Subjects) | Comparator: Placebo (Hispanic Subjects) | Experimental: G-CSF (Black Subjects) | Comparator: Placebo (Black Subjects)
Number analyzed (Participants) | 19 | 21 | 5 | 5 | 6 | 6
Hot flash severity score | -0.29 (0.16) | -0.09 (0.11) | 0.13 (0.14) | -0.13 (0.2) | -0.14 (0.1) | 0.13 (0.21)
Statistical Analysis 1: Comparison: Experimental: G-CSF (White Subjects) vs Comparator: Placebo (White Subjects); Test type: Superiority; p = 0.147, t-test, 1 sided
Statistical Analysis 2: Comparison: Experimental: G-CSF (Hispanic Subjects) vs Comparator: Placebo (Hispanic Subjects); Test type: Superiority; p = 0.160, t-test, 1 sided
Statistical Analysis 3: Comparison: Experimental: G-CSF (Black Subjects) vs Comparator: Placebo (Black Subjects); Test type: Superiority; p = 0.152, t-test, 1 sided

17. Secondary Outcome: Net Change in MENQOL VMS Score
Description: Menopause-specific Quality of Life (MENQOL) Questionnaire. The MENQOL is self-administered and consists of a total of 29 items in a Likert-scale format. Each item assesses the impact of one of four domains of menopausal symptoms, as experienced over the last month: vasomotor (items 1-3), psychosocial (items 4-10), physical (items 11-26), and sexual (items 27-29). MENQOL VMS refers to the answers to items 1-3 where 6 = most bothersome and 0 = least bothersome). (Maximum bothersomeness = 18; No bothersomeness = 0)
Time Frame: Baseline and week 12
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 30 | 29 | 18 | 18
Score on a scale | -5.7 (1.0) | -4.8 (1.2) | -6.0 (1.2) | -3.6 (1.5)
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Test type: Superiority; p = 0.286, t-test, 1 sided
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); Test type: Superiority; p = 0.107, t-test, 1 sided

18. Secondary Outcome: Net Change in HFRDIS Score
Description: The Hot Flash Related Daily Interference Scale (HFRDIS) measures (as a score of 0 to 10) the effect of hot flashes on overall quality of life and on nine specific activities: work, social activities, leisure activities, sleep, mood, concentration, relations with others, sexuality, and enjoyment of life. The 10 answers are added up to get a total score. HFRDIS Score (Maximum Bothersomness = 100; No Bothersomeness = 0). The higher the score, the more bothersome the symptoms.
Time Frame: Baseline and week 12
Population: as for outcome 6
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 28 | 28 | 17 | 18
score on a scale | -22.5 (6.1) | -26.7 (4.5) | -21.2 (7.7) | -25.1 (5.0)
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Test type: Superiority; p = 0.289, t-test, 1 sided
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); Test type: Superiority; p = 0.338, t-test, 1 sided

19. Secondary Outcome: Net Change in ISI Score at 12 Weeks
Description: The Insomnia Severity Index has seven questions. For each question, most bothersome = 4; not bothersome = 0. The seven answers are added up to get a total score. Total score categories: 0-7 = No clinically significant insomnia; 8-14 = Subthreshold insomnia; 15-21 = Clinical insomnia (moderate severity); 22-28 = Clinical insomnia (severe)
Time Frame: Baseline and week 12
Population: as for outcome 6
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 29 | 29 | 17 | 18
score on a scale | -5.5 (1.5) | -6.0 (1.1) | -4.6 (2.0) | -3.8 (1.4)
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Test type: Superiority; p = 0.393, t-test, 1 sided
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); Test type: Superiority; p = 0.365, t-test, 1 sided

20. Secondary Outcome: Net Change in FSS Score at 12 Weeks
Description: Fatigue Severity Scale (FSS) of Sleep Disorders. The Fatigue Severity Scale (FSS) is a method of evaluating the impact of fatigue. The FSS is a short questionnaire (10 questions) that requires the subject to rate level of fatigue. The FSS questionnaire contains nine statements that rate the severity of fatigue symptoms. Each statement is read and the corresponding number from 1 to 7 is circled. A low value (e.g., 1) indicates strong disagreement with the statement, whereas a high value (e.g., 7) indicates strong agreement. (Maximum bother = 70; No bother = 0)
Time Frame: Baseline and week 12
Population: as for outcome 6
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
Number analyzed (Participants) | 28 | 29 | 17 | 18
score on a scale | -5.3 (3.0) | -6.2 (2.2) | -6.9 (3.7) | -7.0 (2.8)
Statistical Analysis 1: Comparison: Experimental: G-CSF (All Subjects) vs Comparator: Placebo/Saline (All Subjects); Test type: Superiority; p = 0.406, t-test, 1 sided
Statistical Analysis 2: Comparison: Experimental: G-CSF (White, NH Subgroup) vs Comparator: Placebo/Saline (White, NH Subgroup); Test type: Superiority; p = 0.494, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: From first dose date up to 30 days after last dose (up to 16 weeks)
Arm/Group | Experimental: G-CSF (All Subjects) | Comparator: Placebo/Saline (All Subjects) | Experimental: G-CSF (White, NH Subgroup) | Comparator: Placebo/Saline (White, NH Subgroup)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 24/30 | 20/30 | 12/18 | 10/18
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: G-CSF (All Subjects) (N=30) | Comparator: Placebo/Saline (All Subjects) (N=30) | Experimental: G-CSF (White, NH Subgroup) (N=18) | Comparator: Placebo/Saline (White, NH Subgroup) (N=18)
General (General disorders) | 10 (10) | 14 (14) | 6 (6) | 7 (7)
Cold/Sinus (Infections and infestations) | 8 (8) | 7 (7) | 4 (4) | 5 (5)
Nausea/GI Disorders (Gastrointestinal disorders) | 4 (4) | 4 (4) | 3 (3) | 0 (0)
Headache (General disorders) | 6 (6) | 1 (1) | 4 (4) | 1 (1)
Fatigue (General disorders) | 6 (6) | 3 (3) | 2 (2) | 2 (2)
Musculo/Skeletal (not incl. bone pain) (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6) | 5 (5) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT03640754/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT03640754/SAP_001.pdf